CLINICAL TRIAL: NCT06960928
Title: Low Dose Sirolimus in People With Post-Acute Sequelae of COVID-19 (PASC) Long COVID-19
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: PolyBio Research Foundation (Other); The Anlyan Center (Unknown)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-24-01366
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Long COVID-19
Keywords: Long COVID-19; Post-Acute Sequelae of COVID-19 (PASC); Sirolimus; Rapamycin
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose sirolimus (Experimental): Participants will follow the escalation scheme and receive sirolimus for up to 12 weeks.
  Interventions: Drug: Low-dose sirolimus
- Placebo (Placebo Comparator): Participants will follow the escalation scheme and receive the placebo for up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose sirolimus — Participants will take sirolimus, at home, for 12 weeks (3 months).
  * 1 pill once a week for 2 weeks (1mg)
  * 2 pills once a week for 2 weeks (2mg)
  * 4 pills once a week for 8 weeks (4mg)
  Other Names: rapamycin
  Arms: Low-dose sirolimus
Drug: Placebo — Participants will take a matching placebo, at home, for 12 weeks (3 months).
  * 1 pill once a week for 2 weeks (0mg)
  * 2 pills once a week for 2 weeks (0mg)
  * 4 pills once a week for 8 weeks (0mg)
  Arms: Placebo

SUMMARY:
The study is conducted in New York, New York at The Cohen Center for Recovery from Complex Chronic Illness at Mount Sinai.

This is an IND-exempt, off-label, multi-ascending, randomized, placebo-controlled clinical trial of sirolimus (also known as rapamycin) in adults with Long COVID. There are 2 arms: Sirolimus and Placebo.

This study aims to evaluate the efficacy of Sirolimus in adults with Long COVID. Efficacy will be evaluated by measuring patient-reported outcomes in response to Sirolimus.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Any sex, aged 18+
* Must be able to attend all study visits located at 5 East 98th St, New York, NY
* Diagnosed with:

  * Long COVID

    * Documented clinical history of confirmed or suspected acute SARS-CoV-2 infection a minimum of 6 months prior to contact with the study team
    * Formal diagnosis of Long COVID from a physician
    * At least a six-month history of one of the following symptoms following SARSCoV-2 infection:

      * headache, memory loss, insomnia, mood disturbance, chest pain, palpitations, shortness of breath, cough, muscle pains, joint pains, or GI upset
      * AND at least moderate fatigue (measured by Fatigue Severity Score)
      * AND at least moderate post-exertional malaise (PEM) (measured by DePaul PEM screener)
      * Participants who are willing and able to comply with all data collection, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
      * Baseline EQ-VAS ≤70; EQ-VAS before the index infection ≥80 (this information is collected before randomization as part of the baseline survey)

Exclusion Criteria:

* Pre-existing conditions including, but not limited to:

  * Autoimmune conditions such as Chronic EBV, Multiple Sclerosis, Hashimoto's Disease, etc. which would impact the immunological profiling analysis.
  * A pre-2020 diagnosis of another Post-Acute Infectious Syndrome such as Chronic Lyme disease, Myalgic Encephalomyelitis/Chronic Fatigue Syndrome, etc.
  * Documented history of vaccine injury
  * History of lung or liver transplant
  * Known hepatic or renal impairment
  * Weighing less than 40 kg
  * Or any other chronic condition that has the potential to impact on immunological profiling, at the discretion of the research physician
* Current use of sirolimus
* Taking a medication with known interactions to sirolimus:

  * Strong CYP3A4 Inhibitors - clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir, such that dose reduction may be necessary
  * Strong CYP3A4 Inducers - carbamazepine, dexamethasone, ethosuximide, glucocorticoids, griseofulvin, phenytoin, primidone, progesterone, rifabutin, rifampin, nafcillin, nelfinavir, nevirapine, oxcarbazepine, phenobarbital, phenylbutazone, rofecoxib (mild), St John's wort, sulfadimidine, sulfinpyrazone, troglitazone, and grapefruit, such that dose increase may be necessary.
  * Drugs that may increase concentration when given with sirolimus - Verapamil, such that dose reduction may be necessary
  * Other drugs that have the potential to increase sirolimus blood concentrations include (but are not limited to): fluconazole, clotrimazole, troleandomycin, nicardipine, cisapride, and metoclopramide
  * Concomitant use of angiotensin-converting enzyme (ACE) inhibitors may increase the risk of developing angioedema.
* Febrile illness within the last 3 months of planned baseline evaluation
* Treatment with another investigational drug or other investigational intervention within 3 months of planned baseline evaluation
* Prophylactic use of aspirin (325 mg daily) for cardiovascular indications will be permitted in participants. All other medications for chronic medical conditions should be initiated at least two months prior to enrollment.
* Uncontrolled diabetes, unstable ischemic heart disease, clinically significant underlying pulmonary disease, history of an immunodeficiency or receiving immunosuppressive therapy; history of coagulopathy or medication condition requiring long-term anticoagulation; history of hepatic impairment; taking angiotensin-converting enzyme (ACE) inhibitors
* Participants who are planning to be or are pregnant
* Participants who are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
European Quality of Life-Visual Analogue Scale (EQ-VAS) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The EQ VAS records the patient's self-rated health on a visual analogue scale where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0), with higher scores indicating better health state. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

SECONDARY OUTCOMES:
The EuroQol Five-Dimensional Health Questionnaire (EQ-5D-5L) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The EQ-5D-5L is a validated, standardized, generic instrument that is a preference-based health- related quality of life questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Full scale from 5 to 25, with higher score indicating poorer health outcomes.
Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. The values of all item responses are averaged to generate subscores for each dimension. From these subscores, a global physical health score and a global mental health score are generated. The scores are translated into T-scores according to a reference population with a mean of 50 and a standard deviation of 10.
General Symptom Questionnaire (GSQ-30) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The General Symptom Questionnaire-30 (GSQ-30) is a valid and reliable instrument to assess symptom burden among patients with acute and post-treatment. The GSQ-30 total score ranges from 0 to 120, with higher scores indicating a greater symptom burden.
Patient Health Questionnaire (PHQ-9) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The PHQ-9 is a series of questions assessing presence and severity of depression symptoms. It evaluates each of the DSM-IV depression criteria and scores the responses from 0 ("Not at all") to 3 ("Nearly every day"). PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively. Full scale from 0-27, with higher score indicating more severe symptoms.
Generalized Anxiety Disorder (GAD-7) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The GAD-7 is a 7-item scale developed and validated to identify generalized anxiety disorder and its severity. It assesses the frequency of 7 anxiety symptoms and scores the responses from 0 ("Not at all") to 3 ("Nearly every day"). Total scores of 5, 10, and 15 correspond to mild, moderate, and severe generalized anxiety disorder, respectively. Full scale from 0-21, with higher score indicating more symptoms.
Neuro-QoL™ v2.0 Cognitive Function-Short Form | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The Neuro-QoL Cognitive Function v2.0 short form assesses perceived difficulties in cognitive abilities, including memory, attention, decision making, planning, organizing, calculating, remembering, and learning. The short form consists of 8 questions assessed on a 5-point Likert scale, resulting in a raw score range of 8 to 40. A raw score is then converted to a T-score using conversion tables. Scores 0.5 - 1.0 SD worse than the mean (T-score 40-45) = mild symptoms/impairment. Scores 1.0 - 2.0 SD worse than the mean (T-score 30-40) = moderate symptoms/impairment. Scores 2.0 SD or more worse than the mean (T-score below 30) = severe symptoms/impairment.
Single-item Sleep Quality Scale (SQS) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)]
  The SQS is a visual analog scale that instructs respondents to rate their overall quality of sleep over a 7-day recall period from 0 to 10. Scores of 0, 1, 4, 7, and 10 correspond to terrible, poor, fair, good, and excellent, respectively. Higher scores indicate better sleep quality.
Fatigue Severity Scale | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The Fatigue Severity Scale (FSS) uses a 7-point scale (1-7) to assess fatigue, with higher scores indicating greater severity, and a total score ranging from 9 to 63. Higher scores indicate more severe fatigue.
Fatigue Visual Analogue Scale [F-VAS]) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The F-VAS consists of 18 items related to fatigue and energy in a visual analogue scale from 0 to 100. A higher score indicates more fatigue.
DePaul Post-Exertional Malaise Questionnaire (DSQ) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The DSQ is designed to evaluate 54 classic ME/CFS symptoms, including fatigue, post-exertional malaise, sleep, pain, neurological/cognitive impairments, and autonomic, neuroendocrine, and immune symptoms. Each symptom's frequency and intensity are rated on a 5-point scale (0-4). Frequency and severity scores are multiplied by 25, added together, and then divided by 2 to create a composite frequency/severity score for each symptom. These scores range from 0 to 100, with higher scores indicating a greater symptom burden.
Composite Autonomic Symptom Score 31(COMPASS-31) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The COMPASS-31 is a 31-question self-assessment instrument of autonomic symptoms and function that is up-to-date, broadly applicable, easy to administer in a short amount of time, and based on a scientific approach. The total score ranges from 0 to 100, with higher scores indicating greater autonomic dysfunction.
Pain (P-VAS) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)]
  Using a visual analogue scale, patients mark a point on a line representing a continuum from "no pain" to "worst pain," with scores ranging from 0 to 100, where higher scores indicate greater pain.
University of California-Los Angeles (UCLA) Loneliness Scale (3-item) | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  The UCLA Loneliness (3-item) Scale scores range from 3 to 9, with higher scores indicating greater perceived loneliness.
Adapted Berkman-Syme Social Network/Connection Index | Baseline (Week 0) and Post-treatment (Week 12 and Week 24)
  This is a self-report questionnaire used to assess social integration and isolation, focusing on marital status, frequency of contact, and participation in social activities, particularly relevant for older adults. Each item is scored on a scale from 1-4 where higher values reflect greater frequency (e.g., 4 = "5 or more times a week"). For each respondent, a sum score is calculated by adding the scores of all five items, yielding a possible score range of 5-25. Higher sum scores reflect higher levels of social connection and lower social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No